CLINICAL TRIAL: NCT03232996
Title: Evaluation of a Computer Game Based Rehabilitation System for Assessment and Treatment of Balance and Gait Impairments in Individuals With Parkinson's Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2017:225
Record Dates: First submitted 2017-07-24; First posted 2017-07-28 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2018-10

CONDITIONS: Parkinson Disease; Parkinson
Keywords: Balance; Gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Computer Game based balance and walk rehabilitation
  Interventions: Other: Computer game based balance and walking rehabilitation for individuals with Parkinson's Disease

INTERVENTIONS:
Other: Computer game based balance and walking rehabilitation for individuals with Parkinson's Disease — All the participants will take part in an 8 week (twice per week) computer game based exercise program for dual task balance and dual task walk training. Participants will be standing in front of LED monitor. They will be asked to wear a head band which will be instrumented with motion sense mouse. Thus, hands-free head rotations will be used to interact with the computer games selected for the DT rehabilitation program. Participants will play few interactive computer games during - Normal standing (fixed surface), Standing on a compliant sponge pad and then while walking on a treadmill.

SUMMARY:
Examining the feasibility and acceptability of the computer game based rehabilitation system for improving balance, gait and executive function in individuals with PD. This will involve a pilot case series intervention study of individuals with PD will be conducted.

DETAILED DESCRIPTION:
This research study will involve a case series pilot study of individuals with PD. Conventional therapy programs for PD population target motor and cognitive deficits in isolation. Recently there has been a growing interest in the application of digital media in rehabilitation. Exergaming and the use of cognitive games have shown good results in patients with Traumatic brain injury, Cerebral palsy, stroke rehabilitation and geriatric population for mobility limitations and dementia.

All the 30 participants from the previous objective will be requested to take part in our objective 2. Objective 2 research protocol will be an 8- week (twice per week) training program of DT balance and DT walking exercises.

Each session will be 45 minutes long. A basic computer game based exercise program will be designed for each participant depending upon their functional status. Every Participant will receive orientation and training about CGBRS, motion mouse and video-games. For initial sessions, relatively slow and large target movements will be selected for the computer games. Game speed, amplitude, mouse sensitivity, and difficulty will be progressed as tolerated for each participant.

Participants will be asked to stand on a stationary treadmill, in front of a LED monitor which will be placed 1 meter away from the treadmill. The treadmill has front and side hand rails so is a convenient place to perform the DT balance activities. The participants will also be fitted with a safety harness. The participants will be asked to wear a head band which is instrumented with the motion sense mouse. Thus, hands-free head rotations will be used to interact with the computer games selected for the DT rehabilitation program. Six to eight computer games will be selected for each participant from a collection of over 60 purchased from Big Fish Games (www.bigfishgames.com). The computer games involve goal-directed visuospatial executive cognitive activities including visual search and tracking of multiple targets, movements of different speeds to interact with game targets with varying movement precision, the presence of distracters, matching and puzzle game.

Participants will play the computer games under the following conditions: -

* While standing on a fixed surface (warm -up duration for 5 minutes)
* While Standing on a compliant sponge pad to increase balance demands (duration - 10 minutes)
* While walking on a treadmill at a predetermined comfortable speed for an interval of 2-3 minutes with 1-2 min rest periods (duration of the treadmill walking component will be 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic PD, defined by the UK Brain Bank criterion
* In disease stage 2 - 3 (classified by Hoehn and Yahr scale)
* Montreal cognitive assessment (MoCA) scores to be 25 or higher
* Able to walk at least 50 meters without any assistance.

Exclusion Criteria:

* Any psychiatric co-morbidity
* Clinically diagnosed dementia or any clinically significant cognitive impairments.
* History of neurological disorder other than PD, which could affect the performance of the participant
* Orthopedic disorders which can affect gait or balance for the participant
* Any unstable medical condition which majorly includes cardiovascular impairments.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Dynamic Standing Balance | Change from baseline Dynamic standing balance at 8 weeks
  The following tasks will be performed for 45 seconds while standing on a sponge pad; a) eyes open (EO), i.e. single task balance condition, and then b) performing the computer gaming activities (i.e. DT balance conditions). A force sensor array (FSA) pressure-sensing mat (Vista Medical Ltd., Manitoba, Canada) will be used to record vertical foot pressures and thus to compute center of foot pressure (COP) migration.
Gait Assessment | Change from baseline spatio-temporal gait variables at 8 weeks.
  The participant will first be asked to walk on the treadmill at his/her comfortable speed for 3 minutes to acclimate with the treadmill prior to testing. After a rest period of 2 minutes they will be asked to walk for 1 minute under the following conditions; a) walk only or single task condition and b) walking while performing the computer gaming tasks (DT walking condition). The treadmill instrumented with a pressure mat (Vista Medical, CA) will be used to record vertical foot contact forces and used to compute spatial-temporal gait variables. Participants walked for 5 minutes to acclimate to the treadmill prior to testing.

SECONDARY OUTCOMES:
Unified Parkinson Disease Rating Scale (UPDRS) | Change from baseline "Final UPDRS scores" at 8 weeks.
  UPDRS is the most common rating scale used to observe and quantify disability and impairment in Parkinson's Disease. This is a 5 point rating scale (from 0 to 5) which is assessed in an ordinal level. 0 describes absence or least severity while 4 describes the highest severity. Increase in severity is denoted with higher scores. Scores will be computed for behavior (part 1), Activites of Daily living (part 2) and Motor (part 3) sections. Scores of all the three section will be added and computed as the "Final UPDRS scores" for our clinical trial

CONTACTS AND LOCATIONS:
Overall Officials: Tony Szturm, Ph.D., Principal Investigator — Professor
Locations (1):
- College of Rehabilitation Sciences, University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bhatt M, Mahana B, Ko JH, Kolesar TA, Kanitkar A, Szturm T. Computerized Dual-Task Testing of Gait Visuomotor and Cognitive Functions in Parkinson's Disease: Test-Retest Reliability and Validity. Front Hum Neurosci. 2021 Jul 15;15:706230. doi: 10.3389/fnhum.2021.706230. eCollection 2021. PMID 34335213